CLINICAL TRIAL: NCT04344639
Title: Incidence, Risk Factors, Severity and Prognosis of Necrotizing Enterocolitis in Turkey: A Prospective Multicentre Study
Brief Title: Incidence, Risk Factors, Severity and Prognosis of Necrotizing Enterocolitis in Turkey
Status: Completed | Type: Observational
Sponsor: Turkish Neonatal Society (Other)
Responsible Party: Principal Investigator, Tolga Hasan Çelik, MD, M.D., Assist. Prof., Division of Neonatology, Department of Pediatrics, Hacettepe University
Other Study IDs: TurkishNECStudyGroup
Record Dates: First submitted 2019-03-05; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Necrotizing Enterocolitis
Keywords: neonate; newborn; premature; necrotizing enterocolitis; neonatal intensive care unit; infant; incidence; risk factors; Turkey
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Risk Factors; Therapeutics; Intensive Care Units, Neonatal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the incidence, risk factors, treatment, prognosis of necrotizing enterocolitis in newborn infants born in newborn intensive care units in our country — With this project, which is planned as a national multicenter prospective study, the incidence of necrotizing enterocolitis in newborn infants born in newborn intensive care units in our country and the risk factors associated with the disease, especially the detailed feeding history of the patient (when the first feeding is nourished, antibiotics and other treatments that are being used). Most epidemiological data such as the most common stage of the disease, treatment, prognosis, comparison with the data of other countries will provide important information for the neonatal health of our country.

SUMMARY:
Necrotizing enterocolitis (NEC) is a gastrointestinal system disease characterized by inflammatory necrosis of the intestine mainly seen in premature infants, and continues to be an important cause of mortality and morbidity in neonatal intensive care units all over the world. Although it is more common in premature infants, it is also seen in term babies when the intestine is ischemic. Although the major problem in premature babies is the immaturity of the intestine, many factors contributing to immaturity play a role in the pathogenesis of NEC.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is a gastrointestinal system disease characterized by inflammatory necrosis of the intestine mainly seen in premature infants, and continues to be an important cause of mortality and morbidity in neonatal intensive care units all over the world. Although it is more common in premature infants, it is also seen in term babies when the intestine is ischemic. Although the major problem in premature babies is the immaturity of the intestine, many factors contributing to immaturity play a role in the pathogenesis of NEC.

With this study project, which is planned as a national multicenter prospective study, the incidence of necrotizing enterocolitis in newborn infants born in neonatal intensive care units in our country and the risk factors associated with the NEC, especially the detailed feeding history of the patient (when the first feeding is nourished, antibiotics and other treatments that are being used). Most epidemiological data such as the most common stage of the disease, treatment, prognosis, comparison with the data of other countries will provide important information for the neonatal health of our country.

The aim of this study was to determine the factors affecting the emergence of NEC in neonatal intensive care units and to determine the frequency of NEC.

Study Hypothesis: Delayed enteral feeding, intensive use of antibiotics and nutrients other than breast milk increase the incidence of necrotizing enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* Newborns diagnosed with NEC in neonatal intensive care units

Exclusion Criteria:

* Major congenital anomaly,
* congenital heart disease (except for atrial septal defect, ventricular septal defect, patent ductus arteriosus)
* Chromosomal anomaly
* Inherited metabolic disease
* Hypoxic ischemic encephalopathy
* Newborns who died within the first 48 hours of life

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns diagnosed with NEC in neonatal intensive care units.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Necrotizing Enterocolitis | 1 year
  Incidence: frequency of NEC during study period
Risk factors for mild and severe necrotizing enterocolitis | 1 year
  erytrocyte/FFP/trombocyte transfusions,PDA closing therapy, umbilical artery catheterisation,
Initiation of enteral feeding time, choice of breastfeeding or formula | 1 year
  nutrition: breastfeeding of formula, delayed enteral feeding
Meconium discharge time | 1 year
  meconium discharge time (hour)
probiotic usage | 1 year
  probiotic usage, type of probiotic preparation
severity of necrotizing enrerocolitis | 1 year
  Grade of NEC disease according to modified Bell Criteria

SECONDARY OUTCOMES:
Prognosis | 1 year
  complications: intestinal perforation, requirement of surgery, short bowell syndrome), mortality rate.

CONTACTS AND LOCATIONS:
Overall Officials: Tolga H Çelik, MD, Principal Investigator — Hacettepe University Faculty of Medicine Department of Pediatrics
Locations (2):
- Turkey (Türkiye) (2):
  - Tolga Hasan Çelik, MD, Ankara
  - Tolga Hasan Çelik, Ankara

IPD SHARING:
Plan to Share IPD: No
This study project is planned as a national multi-center study. This study will be carried out through a Web Based Multicenter Work System, which was formed by the Turkish Neonatal Society.

REFERENCES:
- [Result] Neu J. Necrotizing enterocolitis. World Rev Nutr Diet. 2014;110:253-63. doi: 10.1159/000358474. Epub 2014 Apr 11. PMID 24751635
- [Result] Lim JC, Golden JM, Ford HR. Pathogenesis of neonatal necrotizing enterocolitis. Pediatr Surg Int. 2015 Jun;31(6):509-18. doi: 10.1007/s00383-015-3697-9. Epub 2015 Apr 9. PMID 25854935
- [Result] Kasivajjula H, Maheshwari A. Pathophysiology and current management of necrotizing enterocolitis. Indian J Pediatr. 2014 May;81(5):489-97. doi: 10.1007/s12098-014-1388-5. Epub 2014 Mar 22. PMID 24652270
- [Result] Niemarkt HJ, de Meij TG, van de Velde ME, van der Schee MP, van Goudoever JB, Kramer BW, Andriessen P, de Boer NK. Necrotizing enterocolitis: a clinical review on diagnostic biomarkers and the role of the intestinal microbiota. Inflamm Bowel Dis. 2015 Feb;21(2):436-44. doi: 10.1097/MIB.0000000000000184. PMID 25268636